CLINICAL TRIAL: NCT02153593
Title: Postoperative Bleeding Prevention in Massive Bone Tumour Resection: a Multicentric, Randomized, Parallel, Controlled Trial to Assess the Efficacy of Tranexamic Acid Versus Evicel® and Usual Haemostasis
Brief Title: Postoperative Bleeding Prevention in Massive Bone Tumour Resection
Acronym: TRANEXTUM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-EVI-2011-138; EC11-340 (Other Grant/Funding Number: Ministry of Health and Social Policy 2011); 2011-006276-40 (EudraCT Number)
Record Dates: First submitted 2014-05-27; First posted 2014-06-03 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Blood Loss; Bone Tumour
Keywords: Clinical trial; Randomized; Fibrin glue; Tranexamic acid; Blood loss
MeSH Terms: conditions — Hemorrhage; Bone Neoplasms | interventions — Tranexamic Acid; Fibrin Tissue Adhesive; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranexamic acid (Experimental): Tranexamic acid, 1g intra-articular before closing the surgery wound
  Interventions: Drug: Tranexamic Acid; Procedure: Electrocauterization
- Fibrin glue (Experimental): One intra-articular dose of fibrin glue (Evicel 5mL) before closing the wound surgery
  Interventions: Drug: Fibrin glue; Procedure: Electrocauterization
- Usual hemostasia (Active Comparator): Electrocauterization
  Interventions: Procedure: Electrocauterization

INTERVENTIONS:
Drug: Tranexamic Acid — 1g intra-articular before closing the wound surgery
  Other Names: Amchafibrin
  Arms: Tranexamic acid
Drug: Fibrin glue — 5mL intra-articular before closing the wound surgery
  Other Names: Evicel
  Arms: Fibrin glue
Procedure: Electrocauterization — Coagulation blood from vessels by means of a electrocautery

SUMMARY:
Massive bone tumour resection is often associated with important postoperative bleeding. This may determine systemic (anaemia), as well as local complications (wound healing, seroma, haematoma).

The objective of this study is to determine whether the use of topical tranexamic acid or topical Evicel® will reduce the perioperative bleeding comparing it with usual haemostasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Musculoskeletal tumor (primary or metastatic, benign or malignant) located in extremities, shoulder girdle or pelvis.
* Massive or bloc tumour resection.
* Patient's consent to participate

Exclusion Criteria:

* Known allergy to ATX
* Allergy or known hypersensitivity to bovine proteins (aprotinin)
* Liposarcomas low grade
* History of thromboembolic disease or prothrombotic conditions:

  * cerebral vascular accident
  * ischemic heart disease
  * deep and / or superficial vein thrombosis
  * pulmonary embolism
  * peripheral arterial vasculopathy
  * thrombogenic arrhythmias (eg: ACxFA)
  * patients with cardiovascular stents
  * prothrombotic alterations in coagulation
* Treatment with contraceptive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Total blood loss (mL) in the postoperative period | The first postoperative 48h
  The blood loss will be collected by the drainage system and quantified in mL.

SECONDARY OUTCOMES:
Proportion of patients requiring blood transfusion | The first postoperative 2 weeks
Units of blood transfused | The first postoperative 2 weeks
Proportion of patients with wound infection | The first postoperative month
Proportion of patients with wound dehiscence | The first postoperative month
Proportion of patients with reoperation for wound complications | The first postoperative month
Deep venous thrombosis | The first postoperative 2 weeks
Proportion of patients with seroma | The first postoperative month
Postoperative pain related with the surgery | The first postoperative week
Tumoral local relapse rate | The first postoperative month
Tumoral systemic dissemination rate | The first postoperative month
Mortality | The first postoperative month
Proportion of patients in which chemotherapy is delayed for wound complications | The first postoperative month
Proportion of patients in which radiotherapy is delayed for wound complications. | The first postoperative month
Length of hospital stay | The first postoperative 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ana Peiró, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (3):
- Spain (3):
  - Hospital Universitario de San Juan de Alicante, Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya

REFERENCES:
- [Background] Ibáñez AP, Martinez-Zapata MJ, Tarragó LT, Balaguer MB, Roig XA, Joy IG, Areizaga L, Merino J, Alcalá R, Tranextum Study Group. Postoperative bleeding prevention in massive bone tumour resection: a multicentric, randomized, parallel, controlled trial to assess the efficacy of tranexamic acid versus Evicel and usual haemostasis [protocol]. Basic and Clinical Pharmacology. 2014; 115 (Suppl 3): 20-21.